CLINICAL TRIAL: NCT04181034
Title: Impacts of the Positive Youth Development Program for Expectant and Parenting Teens in California
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Office of Population Affairs (Unknown); California Department of Public Health, MCAH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50023-CA
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Teen Pregnancy Prevention
Keywords: Teen pregnancy prevention; Home visiting; Positive youth development; Adolescent Family Life Program Positive Youth Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PYD (Experimental): Case managers meet with participating pregnant and parenting females at least two times a month over 12 months. In the short term, the program seeks to improve social competence, problem-solving skills, autonomy, increased sense of purpose, improved knowledge and use of contraceptives, increased linkages and support networks, improved quality of relationships, increased access to and strengthen relationship with a trusted adult, increased knowledge of and access to healthcare and improved health and well-being of expectant or parenting mother. In the long term, the program aims to delay subsequent pregnancy and reduction in health risk behaviors, improved health and well-being of parent and child, improved educational and employment outcomes and increased self-sufficiency.
  Interventions: Behavioral: Adolescent Family Life Program Positive Youth Development (PYD) program
- AFLP (Active Comparator): Case managers meet with participating pregnant and parenting females once a month over 24 months to deliver older, business-as-usual version of the program that does not have positive youth development component.
  Interventions: Behavioral: Adolescent Family Life Program (AFLP)

INTERVENTIONS:
Behavioral: Adolescent Family Life Program Positive Youth Development (PYD) program — Home visiting program for pregnant and parenting teens with PYD component
  Arms: PYD
Behavioral: Adolescent Family Life Program (AFLP) — Home visiting program for pregnant and parenting teens
  Arms: AFLP

SUMMARY:
Under contract to the U.S. Department of Health and Human Services (DHHS), Mathematica is conducting an impact study of California Department of Public Health, Center for Family Health, Maternal, Child and Adolescent Health's (MCAH) Adolescent Family Life Program Positive Youth Development (PYD) program for a Federal Evaluation of Programs for Expectant and Parenting Youth (PEPY). The impact study will be designed to address the impact of PYD, compared to the business-as-usual condition, AFLP, in delaying repeat pregnancies, completing high school, improving health of the parent and child, and improving linkages and networks of support for expectant and parenting teens.

DETAILED DESCRIPTION:
The Adolescent Family Life Program (AFLP) has been used by MCAH for more than 3 decades. The program was recently enhanced with a positive youth development component, referred to as Adolescent Family Life Program Positive Youth Development (PYD) program. The enhanced program is a shorter, more intensive program that requires case managers to use motivational interviewing to guide participating youth through a prescribed set of activities designed to set achievable goals for life planning and building self-sufficiency. A random assignment design will be used to assess the program's impact on exposure to program content and short term outcomes.

The evaluation includes two sub-studies, each with a distinct design. In the first sub-study, individuals were randomly assigned as part of the enrollment process within two provider sites to receive either PYD or AFLP. These two provider sites could support individual random assignment because they had enough case managers and clients to support both study conditions (PYD and AFLP). In the second sub-study, 13 provider sites, each with a smaller number of case managers and clients, were randomly assigned to PYD or AFLP. In this second sub-study, participants enrolled after sites were randomly assigned. Potential study participants were recruited between December 2014 and January 2017, and were considered eligible for participation if they were they (1) were interested in the program, (2) were pregnant or parenting, (3) had not been served at the site in the prior six months, (4) spoke either English or Spanish, (5) were between ages 14 and 18, and (6) were not enrolled in Nurse Family Partnerships.

For sub-study 1, potential participants who were eligible were randomly assigned to (1) a treatment group that was eligible for PYD or (2) a control group that received AFLP. Random assignment was conducted within two blocks determined by random assignment site and whether study participants were pregnant at the time of random assignment or were parenting at the time of random assignment. After random assignment, the study enrollment manager assigned the young mother to a case manager delivering the program to which she was assigned. The assigned case manager then tried to locate and conduct a first visit with each randomized youth mother, but not all could be found. For most who were found and visited, case managers were instructed to follow a script that described the program in general terms (without differentiating between AFLP and PYD) and the study in detail. The script did not reveal the group to which the young mother was assigned. As part of the scripted interaction, case managers sought study consent from young mothers to participate in the study data collection.

For sub-study 2, provider sites were first randomized to either the PYD or AFLP. Young mothers were then referred to sites in the same manner as in the first sub-study, went through the same initial eligibility screening process. Eligible mothers were assigned a case manager. The assigned case manager then tried to locate and conduct a first visit with each eligible youth mother, but not all could be found. For most who were found and visited, case managers were instructed to follow a script that described the program in general terms (without differentiating between AFLP and PYD) and the study in detail. The script did not reveal the group to which the young mother was assigned. As part of the scripted interaction, case managers sought study consent from young mothers to participate in the study data collection.

The study draws on data from LodeStar, MCAH's administrative records on service receipt, a baseline survey administered after enrollment into the study, a follow-up survey administered approximately 12 months after enrollment and a follow up survey administered approximately 24 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* must be expectant or parenting

Exclusion Criteria:

* Served by enrollment site in six months prior to random assignment
* Enrolled in Nurse Family Partnership program at time of random assignment
* younger than 14 years of age or older than 18 years of age
* Primary language is neither English nor Spanish

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1330 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Frequency of case manager visits, as measured by administrative data | 12 month
  Continuous variable: Total number of visits with program case manager within the first 12 months from consent date
Frequency of case manager visits, as measured by administrative data | 24 month
  Continuous variable: Total number of visits with program case manager within the first 24 months from consent date
Early exit from program, as measured by administrative data | 12 months
  Binary variable: equal to one if within the first 12 months of programming the participant the participant conveyed the intent to stop programming prematurely to her case manager or became unresponsive to a case manager's attempt to contact.
Exposure to information on relationships in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about relationships, dating, or marriage and that class took place with the case manager or at the recommendation of the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Exposure to information on relationships in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about relationships, dating, or marriage and that class took place with the case manager or at the recommendation of the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on relationships cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about relationships, dating, or marriage and that class took place with the case manager or at the recommendation of the case manager in Year 1 or Year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on parenting in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about parenting or how to care for their child and that class took place with the case manager or at the recommendation of the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Exposure to information on family planning in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable: equal to one if respondent reported receiving information on birth control or where to get birth control from a doctor, nurse, case manager or clinic in Year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Exposure to information on parenting in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about parenting or how to care for their child and that class took place with the case manager or at the recommendation of the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on family planning in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported receiving information on birth control or where to get birth control from a doctor, nurse, case manager or clinic in Year 1, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on parenting cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about parenting or how to care for their child and that class took place with the case manager or at the recommendation of the case manager in Year 1 or Year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on family planning cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable: equal to one if respondent reported receiving information on birth control or where to get birth control from a doctor, nurse, case manager or clinic in Year 1 or Year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on child's access to healthcare in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for their baby or on where to get health care for the their baby addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Exposure to information on child's access to healthcare in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for their baby or on where to get health care for the their baby addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on child's access to healthcare cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for their baby or on where to get health care for the their baby addressed by the case manager directly or through a recommendation by the case manager in Year 1 or Year 2, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to education related services in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: standardized count of education topics addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California". Topics include participating in GED preparation, tutoring, or outside help with school work, or program to prepare for a high school diploma
Exposure to education related services in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of education topics addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include participating in GED preparation, tutoring, or outside help with school work, or program to prepare for a high school diploma
Exposure to education related services cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of education topics addressed by the case manager directly or through a recommendation by the case manager in Years 1 and 2, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include participating in GED preparation, tutoring, or outside help with school work, or program to prepare for a high school diploma
Exposure to workforce assistance related services year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: standardized count of workforce topics addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California". Topics include career counseling, help finding a job or applying for a job training program, job training or help looking for or applying for a job.
Exposure to workforce assistance related services year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of workforce topics addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include career counseling, help finding a job or applying for a job training program, job training or help looking for or applying for a job.
Exposure to workforce assistance related services cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of workforce topics addressed by the case manager directly or through a recommendation by the case manager in year 1 and year 2, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include career counseling, help finding a job or applying for a job training program, job training or help looking for or applying for a job.
Exposure to information on access to healthcare in year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for themselves or on where to get health care for themselves addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Exposure to information on access to healthcare in year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for themselves or on where to get health care for themselves addressed by the case manager directly or through a recommendation by the case manager, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Exposure to information on access to healthcare cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count if respondent reported attending a class or session on how to get health insurance or apply for Medicaid for themselves or on where to get health care for themselves addressed by the case manager directly or through a recommendation by the case manager in year 1 and year 2, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Respondent feelings about themselves, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: proportion of 8 statements related to resiliency & feelings about yourself and the future with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating higher resiliency. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California".
Respondent feelings about themselves, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: proportion of 8 statements related to resiliency & feelings about yourself and the future with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating higher resiliency. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California".
Respondent feelings about personal goals, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: proportion of 7 statements related to resiliency & feelings about personal goals with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating higher resiliency. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California".
Respondent feelings about personal goals, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: proportion of 7 statements related to resiliency & feelings about personal goals with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating higher resiliency. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California".
Linkages and referrals year 1, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: standardized count of topics related to the linkages and referrals addressed by the case manager directly or through a recommendation by the case manager in year 1; variable ranges from 0 to 1, with higher values indicating exposure to more topics about linkages and referrals as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California". Topics include how to get child care for their baby, where to get food assistance and support for themselves and their baby, where to find affordable housing and where to get counseling or treatment for depression or anxiety.
Linkages and referrals year 2, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of topics related to the linkages and referrals addressed by the case manager directly or through a recommendation by the case manager in year 2; variable ranges from 0 to 1, with higher values indicating exposure to more topics about linkages and referrals as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include how to get child care for their baby, where to get food assistance and support for themselves and their baby, where to find affordable housing and where to get counseling or treatment for depression or anxiety.
Linkages and referrals cumulative measure, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: standardized count of topics related to the linkages and referrals addressed by the case manager directly or through a recommendation by the case manager in year 1 and year 2; variable ranges from 0 to 1, with higher values indicating exposure to more topics about linkages and referrals as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California". Topics include how to get child care for their baby, where to get food assistance and support for themselves and their baby, where to find affordable housing and where to get counseling or treatment for depression or anxiety.
Increased access to and strengthened relationship with a trusted adult year 1 | 12 months
  Multiple-item continuous scale variable: Proportion of statements about a supportive adult that the participants agrees with or strongly agrees with, variable ranges from 0 to 1, with higher values indicating more access and stronger relationship with a trusted adult. Each of the four individual statements range from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Increased access to and strengthened relationship with a trusted adult year 2 | 24 months
  Multiple-item continuous scale variable: Proportion of statements about a supportive adult that the participants agrees with or strongly agrees with, variable ranges from 0 to 1, with higher values indicating more access and stronger relationship with a trusted adult. Each of the four individual statements range from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Unprotected sex, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary measure equal to one if the respondent reported having sex without birth control in the three months prior to completing the 12-month survey, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Unprotected sex, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary measure equal to one if the respondent reported having sex without birth control in the three months prior to completing the 24-month survey, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Use of birth control, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary measure equal to one if the respondent indicated currently using condoms, birth control pills, the patch, the shot, the ring, an intrauterine device (IUD) or an implant as a form of birth control, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Use of birth control, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary measure equal to one if the respondent indicated currently using condoms, birth control pills, the patch, the shot, the ring, an intrauterine device (IUD) or an implant as a form of birth control, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Knowledge of condoms, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to six survey items about her knowledge of condoms; each of the six individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Knowledge of condoms, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to six survey items about her knowledge of condoms; each of the six individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Knowledge of birth control pills, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to five survey items about her knowledge of birth control pills; each of the five individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Knowledge of birth control pills, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to five survey items about her knowledge of birth control pills; each of the five individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Knowledge of Intrauterine devices (IUDs), as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to six survey items about her knowledge of IUDs; each of the six individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Knowledge of Intrauterine devices (IUDs), as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to six survey items about her knowledge of IUDs; each of the six individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Knowledge of other hormonal and long-acting reversible contraception (LARC) methods, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to four survey items about her knowledge of other forms of birth control; each of the four individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Knowledge of other hormonal and long-acting reversible contraception (LARC) methods, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable that is the standardized count of the mother's correct responses to four survey items about her knowledge of other forms of birth control; each of the four individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Depressive symptoms, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable equal to one if the respondent was so sad or hopeless for two or more weeks that she stopped doing some usual activities, as measured on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Depressive symptoms, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable equal to one if the respondent was so sad or hopeless for two or more weeks that she stopped doing some usual activities, as measured on the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Received postpartum medical checkup, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable equal to one if the mother reported having a checkup in the 3 months after the child was born, as measured on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Health insurance for respondent, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable equal to one if the respondent reported currently having health insurance , as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Health insurance for respondent, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable equal to one if the respondent reported currently having health insurance , as reported on the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Continued high school attachment, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Binary variable equal to one if the respondent reported being enrolled in high school or having a high school diploma or General Education Diploma (GED) as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"
Continued high school attachment, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable equal to one if the respondent reported being enrolled in high school or having a high school diploma or General Education Diploma (GED) as reported on the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Subsequent pregnancy, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable equal to one if the respondent reported a pregnancy after enrollment in the program as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and/or the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Sexually transmitted disease, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California"and "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Binary variable equal to one if the respondent reported being diagnosed with a sexually transmitted disease after program enrollment as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" and/or the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California"
Positive attitudes towards healthy relationships, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California" | 12 months
  Multiple-item continuous scale variable: proportion of 6 statements related to attitudes towards healthy relationships with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating more positive attitudes toward healthy relationships. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - California".
Positive attitudes towards healthy relationships, as measured by the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California" | 24 months
  Multiple-item continuous scale variable: proportion of 6 statements related to attitudes towards healthy relationships with which the participant either agreed or disagreed, variable ranges from 0 to 1 with higher values indicating more positive attitudes toward healthy relationships. Each of the individual items ranged from 1 to 4 with higher numbers corresponding to stronger agreement. Items collected by using the "Positive Adolescent Futures Final 24 Month Follow-up Survey - California".

CONTACTS AND LOCATIONS:
Overall Officials: Susan Zief, PhD, Principal Investigator — Mathematica Policy Research
Locations (13):
- United States (13):
  - Community Action Partnership of Santa Barbara County, Goleta, California
  - Tiburcio Vasquez Health Center, Hayward, California
  - Lake Family Resource Center, Kelseyville, California
  - AltaMed Health Services, Los Angeles, California
  - El Nido Family Centers, Mission Hills, California
  - Stanislaus County Health Services, Modesto, California
  - Placer County Health and Human Services, Roseville, California
  - Sutter Health Teen Programs, Sacramento, California
  - 1. San Diego Adolescent Pregnancy and Parenting Program (San Diego Unified School District), San Diego, California
  - Felton Institute Family Service Agency of San Francisco, San Francisco, California
  - Planned Parenthood Mar Monte, San Jose, California
  - Community Action Partnership of San Luis Obispo, San Luis Obispo, California
  - Sonoma County Health Department, Santa Rosa, California